CLINICAL TRIAL: NCT02847403
Title: Long-acting Exenatide: a Tool to Stop Cognitive Decline in Dysglycemic Patients With Mild Cognitive Impairment?
Brief Title: Long-acting Exenatide and Cognitive Decline in Dysglycemic Patients
Acronym: DRINN
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Azienda Ospedaliero-Universitaria di Parma (Other)
Responsible Party: Principal Investigator, Alessandra Dei Cas, Research Assistant, MD, PhD, Azienda Ospedaliero-Universitaria di Parma
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015-001850-13
Record Dates: First submitted 2016-07-21; First posted 2016-07-28 (Estimated); Last update posted 2021-08-17 (Actual); Status verified 2021-08

CONDITIONS: Dysglycemia; Cognitive Deficit
Keywords: dysglycemia; MCI; exenatide LAR; GLP-1
MeSH Terms: conditions — Cognition Disorders | interventions — Exenatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- exenatide (Experimental): long-acting exenatide 2 mg subcutaneously once-weekly
  Interventions: Drug: Exenatide
- placebo (Placebo Comparator): no drug assigned
  Interventions: Other: placebo

INTERVENTIONS:
Drug: Exenatide — Patients will be injected subcutaneously 2 mg long-acting exenatide once-weekly. No dose titration is foreseen.
  Other Names: bydureon
  Arms: exenatide
Other: placebo — patients will be seen at the Center for Cognitive Disorders and Dementia according to their usual schedule.
  Arms: placebo

SUMMARY:
The overall objective of the study is to assess the potential effects of the long-acting GLP-1 analogue exenatide in preventing/slowing the progression of cognitive dysfunction and related biomarkers in dysglycemic/prediabetic patients with mild cognitive impairment (MCI).

DETAILED DESCRIPTION:
Type 2 Diabetes Mellitus (T2DM) and Alzheimer's Disease (AD) are two of the most common diseases of aging.The presence of T2DM almost doubles the risk of developing AD and is associated with a faster rate of cognitive decline in those with mild cognitive impairment (MCI). Blood glucose levels are directly associated with accelerated cognitive decline also in subjects with impaired fasting glucose and in individuals without clinical DM. Impaired insulin signaling is critically involved in the natural history of both T2DM and AD and it may represent a common mechanistic link ("common soil") between dysglycemic/prediabetic states and AD development and progression.

The overall objective of the study is to assess the potential effects of the long-acting GLP-1 analogue exenatide in preventing/slowing the progression of cognitive dysfunction and related biomarkers in dysglycemic/prediabetic patients with mild cognitive impairment (MCI).

All eligible patients at V0 will undergo baseline assessments (V1) and will be allocated according to the procedure of randomization to one of the study arms. Follow-up (FU) visits for all subjects will be at 16 (V2) and at 32 weeks (V3) after randomization. Additionally, subjects on active treatment will be admitted weekly to the Outpatient Diabetes Unit of the AOUPR for GLP-1 subcutaneous injections and to check for possible side effects. Subjects in the control arm will be seen at the Center for Dementia (AOUPR) according to their usual schedule.

Laboratory and diagnostic:

At each study visits patients will undergo:

* anthropometric and hemodynamic assessment: weight and height for Body Mass Index (BMI) calculation, waist circumference, ambulatory blood pressure, heart rate;
* blood test collection of metabolic profile: blood collection for metabolic/hormonal profile: fasting plasma glucose, HbA1c, insulin, C-peptide, glucagon, active GLP-1, total gastric inhibitory polypeptide (GIP), total cholesterol, HDL-cholesterol, triglycerides, AST, ALT, pancreatic amylase, lipase, creatinine, eGFR.
* cognitive function tests: ADAS-cog and the quality score of MMSE, Phonemic verbal fluency test; Semantic verbal fluency test; Geriatric Depression Scale (GDS) ; Clinical Dementia Rating Scale (CDR); Neuropsychiatric Inventory (NPI); Activities of Daily Living (ADL); Instrumental Activities of Daily Living (IADL).

ADAS-cog was designed to measure the severity of the most important symptoms of Alzheimer's disease. It consists of 11 7 tasks measuring the disturbances of memory, language, praxis, attention and other cognitive abilities which are often referred to as the core symptoms of AD.

- Functional Magnetic Resonance Imaging (MRI)(only at V1 and V3).

ELIGIBILITY:
Inclusion Criteria:

* patients capable of giving informed consent
* dysglycemia/prediabetes defined as fasting plasma glucose between 100 and 125 mg/dl and/or 2-hour plasma glucose between 140 and 199 mg/dl after a 75 g OGTT and/or a HbA1c value between 5.7 and 6.4%
* diagnosis of MCI according to the Petersen clinical criteria (the expected corrected scores at the MMSE are from 24 to 27)
* age >50<80 yrs
* stable medication for the past 3 months
* Caucasian ethnicity

Exclusion Criteria:

* age <50>80 yrs
* incapability to give informed consent
* diabetes defined according to American Diabetes Association (ADA) criteria
* clinically significant liver or kidney dysfunction defined as s-ALT > 2 times upper reference or estimated creatinine-clearance (eGFR) < 60 mL / min/1.73m2, assessed by with CKD-EPI formula
* endocrinological diseases other than well controlled hypothyroidism, personal or family history of medullary thyroid carcinoma or Multiple Endocrine Neoplasia (MEN) syndrome, severe gastro-intestinal diseases (i.e gastroparesis, dumping syndromes), current or history of chronic or acute pancreatitis
* any contraindication to the use of exenatide as per the Summary of Product Characteristics
* known abuse of alcohol or drugs
* ferro-magnetic prosthesis, pacemaker or other metals incorporated in the body
* significant neurologic disease other than MCI (i.e. Parkinson's disease, multiple system atrophy, normal pressure hydrocephalus, progressive supranuclear palsy, subarachnoid hemorrhage, brain neoplasms, Huntington disease, epilepsy or head trauma)
* BMI ≤22 Kg/m2 in subject ≥ 70 yrs
* MRI/CT showing unambiguous etiological evidence of cerebrovascular disease with regard to MCI
* severe sensory defects; current presence of clinically significant psychiatric disorder
* warfarin treatment, clinically significant systemic condition
* history of cancer within the last 5 yrs
* known allergy to exenatide or any of the other components.

Ages: 51 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-02; Primary Completion 2019-07 (Actual); Study Completion 2021-10-31 (Estimated)

PRIMARY OUTCOMES:
Improvement of ADAS-cog Alzheimer's Disease Assessment Scale defined by ADAS-cog score at 16 (V2) and at 32 weeks (V3) compared to baseline | 16 and 32 weeks
  Absolute difference in the ADAS-Cog score compared to baseline in the 2 arms.

SECONDARY OUTCOMES:
Improvement of Mini Mental State Evaluation test at 16 (V2) and at 32 weeks (V3) compared to baseline | 16 and 32 weeks
  Absolute difference in the Mini Mental State Evaluation (MMSE) score compared to baseline in the 2 arms.
Improvement of Mini Mental State Evaluation quality test at 16 (V2) and at 32 weeks (V3) compared to baseline | 16 and 32 weeks
  Absolute difference in the MMSE quality test score compared to baseline in the 2 arms.
Improvement of Phonemic verbal fluency test at 16 (V2) and at 32 weeks (V3) compared to baseline | 16 and 32 weeks
  Absolute difference in the Phonemic verbal fluency test score compared to baseline in the 2 arms.
Improvement of Semantic verbal fluency test at 16 (V2) and at 32 weeks (V3) compared to baseline | 16 and 32 weeks
  Absolute difference in the Semantic verbal fluency test score compared to baseline in the 2 arms.
Improvement of Geriatric Depression Scale (GDS) test at 16 (V2) and at 32 weeks (V3) compared to baseline | 16 and 32 weeks
  Absolute difference in the GDS test score compared to baseline in the 2 arms.
Improvement of Clinical Dementia Rating Scale (CDR) test at 16 (V2) and at 32 weeks (V3) compared to baseline | 16 and 32 weeks
  Absolute difference in the CDR test score compared to baseline in the 2 arms.
Improvement of Neuropsychiatric Inventory (NPI) test at 16 (V2) and at 32 weeks (V3) compared to baseline | 16 and 32 weeks
  Absolute difference in the NPI test score compared to baseline in the 2 arms.
Improvement of Activities of Daily Living (ADL) test at 16 (V2) and at 32 weeks (V3) compared to baseline | 16 and 32 weeks
  Absolute difference in the ADL test score compared to baseline in the 2 arms.
Improvement of Instrumental Activities of Daily Living (IADL) test at 16 (V2) and at 32 weeks (V3) compared to baseline | 16 and 32 weeks
  Absolute difference in the IADL test score compared to baseline in the 2 arms.
changes in structural and functional connectivity of neural networks as assessed by functional MRI (fMRI) at 16 (V2) and at 32 weeks (V3) | 16 and 32 weeks
  Before and after treatment voxel-wise brain maps will be statistically compared using Statistical Parametric Mapping, by a multivariate 2 x 2 ANOVA (experimental treatment /placebo x time pre/post) in order to observe changes in structural and functional connectivity of neural networks in relation to treatment

CONTACTS AND LOCATIONS:
Overall Officials: Alessandra Dei Cas, MD, Principal Investigator — Azienda Ospedaliero-Universitaria di Parma
Locations (2):
- Italy (2):
  - Endocrinology Unit, Parma
  - Center for Cognitive Disorders and Dementia AUSL of Parma and University of Parma, Parma

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Perry T, Holloway HW, Weerasuriya A, Mouton PR, Duffy K, Mattison JA, Greig NH. Evidence of GLP-1-mediated neuroprotection in an animal model of pyridoxine-induced peripheral sensory neuropathy. Exp Neurol. 2007 Feb;203(2):293-301. doi: 10.1016/j.expneurol.2006.09.028. Epub 2006 Nov 22. PMID 17125767
- [Background] During MJ, Cao L, Zuzga DS, Francis JS, Fitzsimons HL, Jiao X, Bland RJ, Klugmann M, Banks WA, Drucker DJ, Haile CN. Glucagon-like peptide-1 receptor is involved in learning and neuroprotection. Nat Med. 2003 Sep;9(9):1173-9. doi: 10.1038/nm919. Epub 2003 Aug 17. PMID 12925848
- [Background] McClean PL, Holscher C. Liraglutide can reverse memory impairment, synaptic loss and reduce plaque load in aged APP/PS1 mice, a model of Alzheimer's disease. Neuropharmacology. 2014 Jan;76 Pt A:57-67. doi: 10.1016/j.neuropharm.2013.08.005. Epub 2013 Aug 21. PMID 23973293
- [Background] Aviles-Olmos I, Dickson J, Kefalopoulou Z, Djamshidian A, Ell P, Soderlund T, Whitton P, Wyse R, Isaacs T, Lees A, Limousin P, Foltynie T. Exenatide and the treatment of patients with Parkinson's disease. J Clin Invest. 2013 Jun;123(6):2730-6. doi: 10.1172/JCI68295. PMID 23728174